CLINICAL TRIAL: NCT07183280
Title: The Construction and Maintenance of A Real World Study Multicentric Database for Solid Pseudopapillary Neoplasm of the Pancreas
Brief Title: Multicentric Database for Solid Pseudopapillary Neoplasm of the Pancreas
Acronym: SPN
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Prof, Fudan University
Other Study IDs: PTCA199-15
Record Dates: First submitted 2025-09-08; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Solid Pseudopapillary Neoplasm of the Pancreas
Keywords: Solid Pseudopapillary Neoplasm of the Pancreas; Multicenter real-world database
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: operation — Enucleation, spleen-preserving distal pancreatectomy, or duodenum-preserving pancreatic head resection, etc

SUMMARY:
To establish and maintain a reliable multicenter real-world database for pancreatic SPN, providing high-quality data and evidence-based support for clinical/translational research.

DETAILED DESCRIPTION:
Pancreatic solid pseudopapillary neoplasm (SPN) is a low-grade malignant tumor, accounting for 0.2%-2.7% of pancreatic tumors, with unique histological and biological characteristics. Its pathological features include solid-cystic and pseudopapillary structures. SPN occurs predominantly in younger individuals, with a median age of 27-31 years. Male patients tend to be older than female patients, but the incidence is significantly higher in females. This gender disparity may be related to hormonal factors or genetic susceptibility. Although most patients have excellent prognosis (10-year survival rate >95%), approximately 10% may develop metastasis or recurrence, particularly in cases with high-risk pathological features. Reported incidence rates are higher in Asia than in Western countries, with Chinese multicenter studies indicating SPN constitutes 2.8% of pancreatic tumors. SPN exhibits significant differences from other pancreatic tumors in epidemiology, morphology, immunophenotype, and genetics, warranting classification as a distinct pathological entity for clinical management and prognostic evaluation.

Real-world study (RWS) refers to the systematic collection of patient health data in real-world clinical settings [real-world data (RWD)] to address predefined medical questions, employing multidisciplinary methods for comprehensive analysis to generate real-world evidence (RWE). RWS can inform clinical decision-making, support drug development and regulatory decisions, and guide public health policies through pharmacoeconomic evaluations. As an important complement and extension to randomized controlled trials (RCTs), RWS has gained increasing attention globally in recent years. In May 2019, the U.S. FDA issued draft guidance on "Submitting Documents Using Real-World Data and Real-World Evidence to FDA for Drugs and Biologics", detailing the use of RWD/RWE for regulatory approvals. China's NMPA released the "Guideline for Real-World Evidence to Support Drug Development and Evaluation (Trial)" in January 2020, formally incorporating RWE into drug development and regulatory frameworks. Similar initiatives exist in Japan, South Korea, and the EU. As of June 2020, over 2,000 RWS studies were registered globally, including 300+ in China (70+ related to oncology).

SPN is insensitive to chemotherapy and radiotherapy, with complete surgical resection being the cornerstone of cure. R0 resection (negative margins) reduces recurrence and improves survival. For resectable SPN, surgery is strongly recommended. Despite being classified as malignant, SPN exhibits indolent growth with excellent outcomes. Most patients undergoing R0 resection achieve cure. Organ-preserving techniques (e.g., enucleation, spleen-preserving distal pancreatectomy) and minimally invasive approaches (laparoscopic/robotic) are prioritized to reduce complications and enhance quality of life. However, large-scale evidence comparing surgical approaches (minimally invasive vs. open; standard vs. limited resection) remains limited.

Given SPN's rarity and slow research progress, the investigators propose establishing a multicenter RWS database to:

1. Design a tailored database system for SPN, retrospectively collecting clinical data from Shanghai Pancreatic Tumor Institute and other centers;
2. Prospectively collect and maintain SPN patient data to support clinical and translational research.

ELIGIBILITY:
Inclusion Criteria:

* No restrictions on age, gender, or performance status;
* Pathologically/cytologically confirmed SPN;
* Compliance with follow-up requirements;

Exclusion Criteria:

* Non-neoplastic pancreatic lesions;
* Non-pancreatic primary tumors;
* Non-compliance with follow-up;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To establish and maintain a reliable multicenter real-world database for pancreatic SPN, providing high-quality data and evidence-based support for clinical/translational research.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2040-12-30 (Estimated); Study Completion 2041-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 12 month
  OS: OS of subjects from recruiting to the time of death from any cause

SECONDARY OUTCOMES:
Disease free survival (DFS) | up to 10 years
  Disease free survival (DFS) is calculated from completion of surgery and ends when the first event (recurrence/progression/death) occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Luo, Principal Investigator — Shanghai Cancer Center
Locations (1):
- Shanghai Cancer Center, Shanghai, Special Administrative Region, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hua Y, Hong X, Dai M, Li J, Yang S, Guo J, Wang W, Xu Q, Han X, Wang M, Huang N, Zheng H, Kleeff J, Liu Q, Wu W, Zhang T, Liao Q, Zhao Y. Local resection for solid pseudopapillary neoplasms of the pancreas shows improved postoperative gastrointestinal function and reduced mental stress: a multiquestionnaire survey from a large cohort. Int J Surg. 2023 Dec 1;109(12):3815-3826. doi: 10.1097/JS9.0000000000000702. PMID 37830944